CLINICAL TRIAL: NCT00587483
Title: The Use of Amiodarone vs. Lidocaine and Placebo for the Prevention of Ventricular Fibrillation After Myocardial Reperfusion During Cardiopulmonary Bypass
Brief Title: Amiodarone for the Prevention of Reperfusion Ventricular Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: William J. Mauermann, MD, Mayo clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 06-005522; 06-005522 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Results first posted 2011-08-09 (Estimated); Last update posted 2011-08-11 (Estimated); Status verified 2011-07

CONDITIONS: Other Intraoperative Cardiac Functional Disturbances During Cardiac Surgery
Keywords: cardiopulmonary bypass; reperfusion ventricular fibrillation; ventricular fibrillation; amiodarone; lidocaine; cardiac surgery
MeSH Terms: conditions — Ventricular Fibrillation | interventions — Lidocaine; Amiodarone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lidocaine 1.5 mg /kg (Active Comparator): Lidocaine is a class I (sodium channel block) antiarrhythmic drug.
  Interventions: Drug: Lidocaine
- Amiodarone 300 mg (Active Comparator): Amiodarone is used to treat and prevent certain types of serious, life-threatening ventricular arrhythmias (a certain type of abnormal heart rhythm) when other medications did not help or could not be tolerated. Amiodarone is in a class of medications called antiarrhythmics. It works by relaxing overactive heart muscles.
  Interventions: Drug: Amiodarone
- placebo (saline) (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lidocaine — Lidocaine is a class I (sodium channel block) antiarrhythmic drug
  Other Names: lidocaine cardioplegia; Xylocaine; lidocaine hydrochloride
  Arms: Lidocaine 1.5 mg /kg
Drug: Amiodarone — 300 mg
  Other Names: Cordarone; Pacerone
  Arms: Amiodarone 300 mg
Drug: Placebo — Saline
  Arms: placebo (saline)

SUMMARY:
This was a prospective, randomized, double blinded study in which patients undergoing a cardiopulmonary bypass (CPB) with aortic cross clamping were randomly assigned to receive amiodarone, lidocaine, or saline placebo prior to removal of the aortic cross clamp. (CPB is a technique that temporarily takes over the function of the heart and lungs during surgery, maintaining the circulation of blood and the oxygen content of the body.) Specifically, we will test the hypothesis that amiodarone is superior to both lidocaine and placebo in the prevention of a severely abnormal heart rhythm when the blood flow is restored to the heart after the aortic cross clamp is removed.

DETAILED DESCRIPTION:
This was a prospective, randomized, double blinded study in which patients undergoing cardiopulmonary bypass with aortic cross clamping were randomly assigned to receive amiodarone, lidocaine, or saline placebo prior to removal of the aortic cross clamp. Specifically, we will test the hypothesis that amiodarone administration decreases the incidence of ventricular fibrillation, the number of defibrillation attempts and the total energy and current required for defibrillation should ventricular fibrillation occur.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cardiac surgery that was expected to include cross-clamping of the aorta

Exclusion Criteria:

* Women wishing to become pregnant within 6 months of surgery
* Allergy to amiodarone
* History of organ dysfunction due to previous amiodarone use
* Patients who require more than mild systemic hypothermia (<32 degrees C) during cardiopulmonary bypass
* Patients who require more than one bypass run or more than one period of aortic cross-clamping

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342 (Actual)
Dates: Start 2007-11; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William J Mauermann, MD, Principal Investigator — clinical instructor
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Mauermann WJ, Pulido JN, Barbara DW, Abel MD, Li Z, Meade LA, Schaff HV, White RD. Amiodarone versus lidocaine and placebo for the prevention of ventricular fibrillation after aortic crossclamping: a randomized, double-blind, placebo-controlled trial. J Thorac Cardiovasc Surg. 2012 Nov;144(5):1229-34. doi: 10.1016/j.jtcvs.2012.06.039. Epub 2012 Jul 4. PMID 22770549

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult patients presenting for cardiac surgery in which aortic cross clamping was anticipated were recruited between 11/2007 and 6/2010
Groups:
- Lidocaine 1.5 mg /kg: Subjects randomized to receive Lidocaine 1.5 mg/kg via the cardiopulmonary reservoir prior to the removal of the aortic cross clamp.
- Amiodarone 300 mg: Subjects randomized to receive Amiodarone 300 mg IV(followed by 150 mg IV if needed) via the cardiopulmonary reservoir prior to the removal of the aortic cross clamp.
- Placebo (Saline): Subjects randomized to receive placebo (saline) via the cardiopulmonary reservoir prior to the removal of the aortic cross clamp.
Period: Overall Study
Arm/Group | Lidocaine 1.5 mg /kg | Amiodarone 300 mg | Placebo (Saline)
Started | 115 | 115 | 112
Completed | 115 | 115 | 112
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lidocaine 1.5 mg /kg | Amiodarone 300 mg | Placebo (Saline) | Total
Number analyzed (Participants) | 115 | 115 | 112 | 342
Age Continuous [Mean (Standard Deviation); unit: years] | 62.7 (13.9) | 63.3 (13.6) | 63.6 (13.0) | 63.2 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 41 | 30 | 105
  Male | 81 | 74 | 82 | 237
Type of Operation [Number; unit: Participants] — The planned operative procedure requiring cardiopulmonary bypass with aortic cross clamping.
  Participants
    Coronary Artery Bypass Grafting only | 15 | 18 | 20 | 53
    Valve only | 37 | 38 | 31 | 106
    Septal Myectomy | 30 | 34 | 34 | 98
    Multiple Procedures | 33 | 25 | 27 | 85
Preoperative Medications [Number; unit: Participants] — Participants could have received more than one preoperative medication, therefore the totals of all the medications are greater than the number of participants.
  Participants
    Beta blocker | 73 | 67 | 73 | 213
    ACE Inhibitor/Angiotensin Receptor Blocker (ARB) | 31 | 43 | 29 | 103
    Statin | 42 | 46 | 60 | 148
    Digoxin | 4 | 7 | 7 | 18
    Amiodarone | 7 | 5 | 2 | 14
History of Dysrhythmias [Number; unit: Participants]
  Atrial Fibrillation | 22 | 23 | 17 | 62
  Atrial Flutter | 2 | 4 | 1 | 7
  Ventricular | 3 | 0 | 3 | 6
  Unknown or Not Reported | 88 | 88 | 91 | 267
Left Ventricular Ejection Fraction (%) [Mean (Standard Deviation); unit: Percentage] | 62.7 (11.5) | 62.7 (10.8) | 62.8 (11.7) | 62.75 (11)
Medical History/Comorbidities [Number; unit: Participants] — Participants could have had more than one pre-existing condition, therefore the totals may be greater or less than the total number of participants in each group.
  Participants
    Diabetes Mellitus | 14 | 16 | 14 | 44
    Chronic Obstructive Pulmonary Disease (COPD) | 7 | 3 | 5 | 15
    Hypertension | 37 | 55 | 48 | 140
    Unknown or Not Reported | 57 | 41 | 45 | 143

OUTCOME MEASURES:

1. Primary Outcome: Participants Experiencing Ventricular Fibrillation Requiring Defibrillation During the 60 Minute Period Following Myocardial Reperfusion
Time Frame: Participants were followed from randomization through the 60 minute period following myocardial reperfusion.
Population: Intention to Treat (ITT)
Measure: Number; unit: Participants
Arm/Group | Lidocaine 1.5 mg /kg | Amiodarone 300 mg | Placebo (Saline)
Number analyzed (Participants) | 115 | 115 | 112
Participants | 66 | 60 | 70
Statistical Analysis 1: Comparison: Lidocaine 1.5 mg /kg vs Amiodarone 300 mg; The expected overall incidence of ventricular fibrillation after removal of the aortic clamp is at least 70%. Using a chi square analysis with 80% power and an alpha of 0.0167, we estimate that we will need 113 patients in each group to show a 30% reduction in the incidence of ventricular fibrillation with amiodarone; Test type: Superiority or Other; p = 0.427, Regression, Logistic — An alpha of 0.0167 was used to account for multiple comparisons among the 3 groups. Given the total of 3 comparisons, 0.05/3 = 0.0167 was used in the calculation; Odds Ratio (OR) = 0.81, 95% CI 2-sided [0.48 to 1.37]
Statistical Analysis 2: Comparison: Amiodarone 300 mg vs Placebo (Saline); Test type: Superiority or Other; p = 0.117, Regression, Logistic; Odds Ratio (OR) = 0.65, 95% CI 2-sided [0.39 to 1.11]
Statistical Analysis 3: Comparison: Lidocaine 1.5 mg /kg vs Placebo (Saline); Test type: Superiority or Other; p = 0.433, Regression, Logistic; Odds Ratio (OR) = 0.80, 95% CI 2-sided [0.47 to 1.37]

2. Secondary Outcome: Number of Defibrillation Attempts
Time Frame: Participants were followed from randomization through the 60 minute period following myocardial reperfusion.
Population: Intention to Treat (IIT)
Measure: Number; unit: Participants
Arm/Group | Lidocaine 1.5 mg /kg | Amiodarone 300 mg | Placebo (Saline)
Number analyzed (Participants) | 115 | 115 | 112
Participants
  0 Attempts | 46 | 57 | 40
  1 - 3 Attempts | 53 | 43 | 46
  > 3 Attempts | 16 | 15 | 14
Statistical Analysis 1: Comparison: Lidocaine 1.5 mg /kg vs Amiodarone 300 mg; Test type: Superiority or Other; p = 0.215, Regression, Logistic; Odds Ratio (OR) = 0.74, 95% CI 2-sided [0.45 to 1.19]
Statistical Analysis 2: Comparison: Amiodarone 300 mg vs Placebo (Saline); Test type: Superiority or Other; p = 0.008, Regression, Logistic; Odds Ratio (OR) = 0.51, 95% CI 2-sided [0.32 to 0.84]
Statistical Analysis 3: Comparison: Lidocaine 1.5 mg /kg vs Placebo (Saline); Test type: Superiority or Other; p = 0.424, Regression, Logistic; Odds Ratio (OR) = 0.82, 95% CI 2-sided [0.52 to 1.33]

3. Secondary Outcome: Incidence of Arrhythmias Other Than Ventricular Fibrillation
Description: Number of participants per arm who experienced arrhythmias other than ventricular fibrillation while in the ICU.
Time Frame: Participants were followed from randomization through the 60 minute period following myocardial reperfusion.
Measure: Number; unit: Participants
Arm/Group | Lidocaine 1.5 mg /kg | Amiodarone 300 mg | Placebo (Saline)
Number analyzed (Participants) | 115 | 114 | 111
Participants
  Ventricular tachycardia | 3 | 2 | 0
  Atrial fibrillation | 21 | 23 | 18
  Other arrhythmias | 27 | 35 | 27

4. Secondary Outcome: Incidence of Arrhythmias in the Post-Operative Period
Description: Number of participants per arm who experienced arrhythmias while on floor care following dismissal from the ICU.
Time Frame: Participants were followed from dismissal from the ICU until dismissal from the hospital.
Measure: Number; unit: Participants
Arm/Group | Lidocaine 1.5 mg /kg | Amiodarone 300 mg | Placebo (Saline)
Number analyzed (Participants) | 115 | 114 | 111
Participants
  Ventricular tachycardia | 2 | 2 | 3
  Atrial fibrillation | 56 | 49 | 38
  Other arrhythmias | 36 | 42 | 24

5. Secondary Outcome: Use of Vasopressors
Description: Number of participants per arm who required the use of vasopressors in the post-operative period.
Time Frame: Participants were followed from randomization until time to discharge from the hospital.
Measure: Number; unit: Participants
Arm/Group | Lidocaine 1.5 mg /kg | Amiodarone 300 mg | Placebo (Saline)
Number analyzed (Participants) | 115 | 114 | 111
Participants
  Epinephrine | 1 | 1 | 0
  Norepinephrine | 0 | 0 | 0
  Vasopressin | 0 | 2 | 0

6. Secondary Outcome: Time to Discharge From the Intensive Care Unit
Time Frame: Participants were followed from the date of randomization until the date of discharge from the Intensive Care Unit, assessed up to 40 days.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Lidocaine 1.5 mg /kg | Amiodarone 300 mg | Placebo (Saline)
Number analyzed (Participants) | 115 | 114 | 111
Days | 1.357 (0.948) | 5.329 (34.515) | 4.847 (34.622)

7. Secondary Outcome: Time to Discharge From the Hospital
Time Frame: Participants were followed from the date of randomization until the date of discharge from the hospital, assessed up to 60 days.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Lidocaine 1.5 mg /kg | Amiodarone 300 mg | Placebo (Saline)
Number analyzed (Participants) | 115 | 114 | 111
Days | 6.183 (2.833) | 7.5 (8.545) | 9.423 (34.572)

ADVERSE EVENTS:
Arm/Group | Lidocaine 1.5 mg /kg | Amiodarone 300 mg | Placebo (Saline)
Serious Adverse Events (participants affected / at risk) | 0/115 | 0/115 | 0/112
Other Adverse Events (participants affected / at risk) | 0/115 | 0/115 | 0/112

LIMITATIONS AND CAVEATS:
Included a heterogeneous group of operations which possibly make our results applicable to "real world" perioperative care; dosing of amiodarone was higher than in previous investigations, but the dose may not have been large enough.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes